CLINICAL TRIAL: NCT02654158
Title: Phase IV Trial,The Efficacy and Safety Study of Fuganlin Oral Liquid in Children With Acute Upper Respiratory Infection
Status: Completed | Type: Observational
Sponsor: Guangzhou Yipinhong Pharmaceutical CO.,LTD (Industry)
Responsible Party: Sponsor
Other Study IDs: 2013Pro234.EKZY
Record Dates: First submitted 2016-01-11; First posted 2016-01-13 (Estimated); Last update posted 2017-05-22 (Actual); Status verified 2016-01

CONDITIONS: Acute Upper Respiratory Infection
Keywords: acute upper respiratory infection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Low-dose of Fuganlin Oral Liquid: oral
  less than 1 years old: 5mL each time and three times a day
  1~3 years old: 10mL each time and three times a day
  4~6 years old: 10mL each time and four times a day
  7~12 years old: 10mL each time and five times a day
  Interventions: Drug: Low-dose of Fuganlin Oral Liquid
- High-dose of Fuganlin Oral Liquid: oral
  less than 1 years old: 10mL each time and three times a day
  1~3 years old: 20mL each time and three times a day
  4~6 years old: 20mL each time and four times a day
  7~12 years old: 20mL each time and five times a day
  Interventions: Drug: High-dose of Fuganlin Oral Liquid

INTERVENTIONS:
Drug: Low-dose of Fuganlin Oral Liquid — less than 1 years old: 5mL each time and three times a day
  1~3 years old: 10mL each time and three times a day
  4~6 years old: 10mL each time and four times a day
  7~12 years old: 10mL each time and five times a day
  Other Names: No other names
  Groups: Low-dose of Fuganlin Oral Liquid
Drug: High-dose of Fuganlin Oral Liquid — less than 1 years old: 10mL each time and three times a day
  1~3 years old: 20mL each time and three times a day
  4~6 years old: 20mL each time and four times a day
  7~12 years old: 20mL each time and five times a day
  Other Names: No other names
  Groups: High-dose of Fuganlin Oral Liquid

SUMMARY:
Phase IV trial,Single-arm, multi-centre clinical trial to assess the efficacy and safety of Fuganlin Oral Liquid in children with acute upper respiratory infection

DETAILED DESCRIPTION:
Low-dose group of Fuganlin Oral Liquid:dosage from 5 to 10 ml;

High-dose group of Fuganlin Oral Liquid:dosage from 10 to 20 ml;

Treatment for 1 week.Patients who were recovered within 1 week can withdrawal at any time.

Research purpose:

1. Evaluate the safety and efficacy of Fuganlin oral Liquid when expanding the designated indications(Qi deficiency wind-heat syndrome to wind-heat syndrome) .
2. Explore the relationship between elevated white blood cells and efficacy, age and efficacy, dose and efficacy,While treating with Fuganlin oral Liquid in children with acute respiratory infection.
3. Observe the antiviral and immunomodulatory effects of Fuganlin oral Liquid.
4. Provide data to support the clinical medicine guidelines and labels amendment of Fuganlin oral Liquid.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed as acute upper respiratory infection.
2. Patients with acute upper respiratory infection diagnosed as Tradition Chinese Medicine syndrome qi deficiency wind-heat.
3. Patients aged 1 to 12 years old.
4. Parents or guardians agreed to participate this study and signed the informed consent.

Exclusion Criteria:

1. Patients whose total numbers of white blood cells around above1.3ULN.
2. Patients diagnosed as suppurative tonsillitis, otitis media, bronchitis and other airway.
3. Patients allergic to the test drug.
4. Serious cardiovascular, liver,kidney and other primary systemic diseases.
5. Patients should not be included in group according to investigator's evaluation.

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children aged 1 to 12 years old with acute upper respiratory infection
Sampling Method: Probability Sample
Enrollment: 2400 (Actual)
Dates: Start 2013-08; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Duration of cold symptoms | Defined as the time from the onset of the cold to the time achieve a cold cure standard,time average 1 to 7 days
  Cold diagnostic criteria：
  1. Nasal congestion, runny nose, sneezing, itchy throat, or pain, cough
  2. The chills, fever, no sweat or less sweat, headache, limb sour
  3. The total numbers of normal or low white blood cells, neutropenia, relative increase in lymphocytes.
  Cold cure criteria:
  1. Fever, aversion to wind individual symptoms disappeared
  2. Nasal congestion, runny nose, sore throat, cough individual symptoms disappeared

CONTACTS AND LOCATIONS:
Overall Officials: Li xinmin, PhD, Study Chair — The First Affiliated Hospital of Tianjing University of Traditional Chinese Medicine; Chang ke, MD, Principal Investigator — Chengdu University of Traditional Chinese Medicine; Meng qingping, MD, Principal Investigator — Zhengzhou Children's Hospital; Tao lei, MD, Principal Investigator — Huanggang Maternal and Child Health Hospital; Ding ying, MD, Principal Investigator — Children's Hospital of The First Affiliated Hospital of Henan College of Traditional Chinese Medicine; Xiang xixiong, PhD, Principal Investigator — Hubei Hospital of Traditional Chinese Medicine; Cheng ji, MD, Principal Investigator — Second Affiliated Hospital of Wenzhou Medical University; Ying yong, MD, Principal Investigator — Affiliated Shanghai Children's Medical Center of Shanghai Jiaotong University School of medicine; Liu changshan, MD, Principal Investigator — Tianjin Medical University Second Hospital; Mou qinghui, MD, Principal Investigator — Jinan children's hospital; Liu yulin, MD, Principal Investigator — BoAi Hospital of Zhongshan; Wang lisheng, PhD, Principal Investigator — Shenzhen Children's Hospital; Zhao deyu, PhD, Principal Investigator — Affiliated Nanjing Children's Hospital of Nanjing Medical University; Du yonggang, MD, Principal Investigator — Changzhi People's Hospital; Su baoling, MD, Principal Investigator — Affiliated Heji Hospital of Changzhi Medical College; Qing yanhong, MD, Principal Investigator — Affiliated Hospital of Shanxi College of Traditional Chinese medicine; Cheng zhimin, PhD, Principal Investigator — Affiliated Children's Hospital of Zhejiang University School of Medicine; Lin yan, MD, Principal Investigator — Chengdu Women and Children's Hospital; Xu youjia, MD, Principal Investigator — Guangdong Provincial Hospital of Traditional Chinese Medicine; Zhang mingying, MD, Principal Investigator — Beijing Shunyi Hospital of China Medical University
Locations (1):
- Guangdong Provincial Hospital of Traditional Chinese Medicine, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided